CLINICAL TRIAL: NCT04029493
Title: The Situation of Re-infection of Helicobacter Pylori After Successful Eradication
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Other Study IDs: 2018SDU-QILU-G116
Record Dates: First submitted 2019-07-21; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Helicobacter Pylori
Keywords: Re-infection
MeSH Terms: conditions — Reinfection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The patients who accept the quadruple eradication program of the helicobacter pylori and success to eradicate helicobacter pylori will be followed-up to observe the situation of re-infection of helicobacter pylori.

DETAILED DESCRIPTION:
The patients with helicobacter pylori accepted he quadruple eradication program of the helicobacter pylori.They will be followed-up from 1 year to 5 years to observe the situation of re-infection of helicobacter pylori.The rate of the re-infection will be described by frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged between 18 and 70 years old, with positive H. pylori infection that was not eradicated by previous therapies are included. The H. pylori infection is confirmed by the positive rapid urease test or 13C-breath test.

Exclusion Criteria:

* Patients with significant underlying disease including liver, cardiac, pulmonary, and renal diseases, neoplasia, coagulopathy and genetic diseases, history of gastric surgery, pregnancy, breast-feeding, active gastrointestinal bleeding, the use of PPI, NSAID or antibiotics during the 4 weeks prior to enrolment, and previous history of allergic reactions to any of the medications used in this protocol. Patients previously treated with H. pylori eradication regimens or those unwilling to participate in the study were also excluded.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The patients in Shandong province, aged between 18 and 70 years old, with previous positive H. pylori infection that suceessed to be eradicated by therapies are included.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The rate of re-infection | 4 years
  The rate of re-infection will be described by the frequency and percentage.

SECONDARY OUTCOMES:
The influence factors of the rate of re-infection | 4 years
  The chi-square test will be used to compare the influence factors of the rate of re-infection.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Study Chair — Qilu Hospital of Shandong University; Tian Ma, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided